CLINICAL TRIAL: NCT04739046
Title: A Single Arm, Open, Exploratory Clinical Trial to Evaluate Efficacy and Safety for Combination Treatment of Replication Competent Adenovirus Double Suicide Gene Therapy(Theragene®,Ad5-yCD/mutTKSR39rep-ADP) and Radiation Therapy in Patients
Brief Title: An Exploratory Trial to Evaluate Efficacy and Safety for Combination Treatment of Adenovirus Double Suicide Gene Therapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: NewGenPharm Incoporation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNUBH-IMGPB-2021-02
Record Dates: First submitted 2021-02-01; First posted 2021-02-04 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-01

CONDITIONS: Pancreas Cancer
Keywords: pancreatic cancer; radiation therapy; adenovirus; gene therapy
MeSH Terms: conditions — Pancreatic Neoplasms; Adenoviridae Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Theragene arm (Experimental): Patients who were treated with Theragene®,Ad5-yCD/mutTKSR39rep-ADP and radiation therapy
  Interventions: Drug: Theragene arm

INTERVENTIONS:
Drug: Theragene arm — Theragene®,Ad5-yCD/ mutTKSR39rep-ADP with radiation therapy

SUMMARY:
Replication-competent Adenovirus-mediated Double Suicide Gene Therapy (Theragene®,Ad5-yCD/mutTKSR39rep-ADP) showed safety and anti-cancer effect in patients with pancreatic cancer in phase I study.

From the experience of phase I study, the safety and efficacy of combination with standard chemotherapy and radiation therapy with Theragene treatment will be assessed in this study.

DETAILED DESCRIPTION:
Phase IIa study of Replication-competent Adenovirus-mediated Double Suicide Gene Therapy (Theragene®,Ad5-yCD/mutTKSR39rep-ADP) with radiation therapy

ELIGIBILITY:
Inclusion Criteria:

* Patients with borderline resectable or locally advanced pancreatic cancer
* Patients with histologically confirmed pancreatic adenocarcinoma
* Patients with no evidence of peritoneal or hematogenous metastasis
* Patients with ECOG performance status 0-1
* Patients with renal function (Serum creatinine ≤ 1.5 mg/dL or creatinine clearance ≥ 50 mL/min/m²)
* Patients with bone marrow function (WBC > 4,000/uL or absolute neutrophil count ≥ 1500/uL, PLT ≥ 100,000/uL, and Hemoglobin > 10 g/dL)
* Patients with liver function (Bilirubin < 2.0 mg/dL and SGOT and SGPT < 3 times upper limit of normal (ULN))
* Patients with agreement with informed consent

Exclusion Criteria:

* Patients with a history of other cancer
* Patients with recurred pancreatic cancer
* Patients with a history of radiation on more than 25% of bone marrow
* Patients with a history of major surgery except laparoscopic examination, endoscopic intervention, or gastrojejunostomy
* Patients who have contraindication of radiation therapy
* Patients with HIV infection, chronic hepatitis B, chronic hepatitis C, or liver cirrhosis
* Female patients with childbearing age or pregnancy or breast feeding
* Patients who are considered as inappropriate candidate by investigators

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 24 weeks
  the proportion of patients with advanced or metastatic cancer who have achieved complete response or partial response

SECONDARY OUTCOMES:
Disease control rate | 24 weeks
  the proportion of patients with advanced or metastatic cancer who have achieved complete response, partial response or stable disease
Tumor marker test | 24 weeks
  change of tumor marker in the process of assigned treatment
Overall survival | 2 years
  median time from beginning of treatment to death

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Hyeok Hwang, MD PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea